CLINICAL TRIAL: NCT06692647
Title: A Two-period Study to Evaluate the Effects of Multiple Oral Doses of Diltiazem on the Single-dose Pharmacokinetics of MK-4318 in Healthy Participants
Brief Title: A Clinical Study of MK-4318 and Diltiazem in Healthy People (MK-4318-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4318-003; MK-4318-003 (Other: MSD)
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Pain
MeSH Terms: conditions — Pain | interventions — Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-4318 Plus Diltiazem (Experimental): Participants will move sequentially through 2 Periods. In Period 1, participants receive MK-4318 orally. In Period 2, participants receive MK-4318 orally plus diltiazem orally.
  Interventions: Drug: MK-4318; Drug: Diltiazem

INTERVENTIONS:
Drug: MK-4318 — Oral administration
Drug: Diltiazem — Oral administration
  Other Names: Cardizem®; Cartia XT®; Matzim LA®

SUMMARY:
The goal of this study is to learn what happens to MK-4318 in a person's body over time. Researchers will compare what happens to levels of MK-4318 in people's blood when it is taken with and without diltiazem. Researchers also want to learn about the safety of MK-4318 taken with and without diltiazem and if people tolerate them.

ELIGIBILITY:
Inclusion Criteria

The main inclusion criteria include but are not limited to the following:

* Is in good health based on medical history and physical examination
* Has a body mass index >18 and ≤32 kg/m^2, inclusive

Exclusion Criteria

The main exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cardiac arrythmia or recurrent unexplained syncopal events

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) of MK-4318 | At designated timepoints (up to approximately 4 days postdose)
  Blood samples will be collected to determine the AUC0-inf of MK-4318 in the presence of diltiazem.
Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24hrs) of MK-4318 | At designated timepoints (up to approximately 1 day postdose)
  Blood samples will be collected to determine the AUC0-24hrs of MK-4318 in the presence of diltiazem.
Plasma Concentration of MK-4318 at 12 Hours Postdose (C12hrs) | At designated timepoints (up to approximately 12 hours postdose)
  Blood samples will be collected to determine the C12hrs of MK-4318 in the presence of diltiazem.
Plasma Concentration of MK-4318 at 24 Hours Postdose (C24hrs) | At designated timepoints (up to approximately 1 day postdose)
  Blood samples will be collected to determine the C24hrs of MK-4318 in the presence of diltiazem.
Maximum Plasma Concentration (Cmax) of MK-4318 | At designated timepoints (up to approximately 4 days postdose)
  Blood samples will be collected to determine the Cmax of MK-4318 in the presence of diltiazem.
Time to Maximum Plasma Concentration (Tmax) of MK-4318 | At designated timepoints (up to approximately 4 days postdose)
  Blood samples will be collected to determine the Tmax of MK-4318 in the presence of diltiazem.
Apparent Clearance (CL/F) of MK-4318 | At designated timepoints (up to approximately 4 days postdose)
  Blood samples will be collected to determine the CL/F of MK-4318 in the presence of diltiazem.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of MK-4318 | At designated timepoints (up to approximately 4 days postdose)
  Blood samples will be collected to determine the Vz/F of MK-4318 in the presence of diltiazem.
Apparent Terminal Half-life (t1/2) of MK-4318 | At designated timepoints (up to approximately 4 days postdose)
  Blood samples will be collected to determine the t1/2 of MK-4318 in the presence of diltiazem.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 60 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Intervention Due to an AE | Up to approximately 9 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study intervention due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Labcorb CRU, Madison (Site 0001), Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com